CLINICAL TRIAL: NCT03717467
Title: The Influence of Intraoperative Magnesium Sulfate Administration on Postoperative Morphine Requirement in Living Donor During Orthotopic Liver Transplantation
Brief Title: Intraoperative Magnesium Sulfate Administration During Orthotopic Liver Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Hany M Yassin, MD, Associate professor of anesthesia, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: D129
Record Dates: First submitted 2018-10-22; First posted 2018-10-24 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Postoperative Pain
Keywords: Magnesium sulfate; Morphine requirement; Hepatotomy; Orthotopic liver transplantation
MeSH Terms: conditions — Pain, Postoperative | interventions — Sodium Chloride; Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patient will be randomly assigned to one of the two groups. An independent anesthesiologist who will not be participating in the study prepares the study medications.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S group (Placebo Comparator): Isotonic saline as placebo will be given.
  Interventions: Drug: isotonic saline
- M group (Active Comparator): Magnesium sulfate will be given
  Interventions: Drug: Magnesium Sulfate

INTERVENTIONS:
Drug: isotonic saline — 100 ml of isotonic saline over 15 min immediately before induction of anesthesia and then 15 mg/kg/h by continuous I.V. infusion until the end of operation.
  Other Names: Saline group
  Arms: S group
Drug: Magnesium Sulfate — 40 mg/kg of magnesium sulfate in 100 ml of isotonic saline over 15 min immediately before induction of anesthesia and then 15 mg/kg/h by continuous I.V. infusion until the end of operation.
  Other Names: Magnesium group
  Arms: M group

SUMMARY:
The aim of study is to assess the effect of intraoperative use of magnesium sulfate in liver donating patients in reducing post-operative morphine requirements in early postoperative 24 hour in adult living liver donor.The authors hypothesize that magnesium sulfate can be used to efficiently reduce postoperative morphine consumption in the early 24 hours postoperatively as evident in other surgery types.

DETAILED DESCRIPTION:
Introduction A lot of recent trials emphasized that perioperative magnesium sulfate (MgSO4) infusion has general anesthetic properties that could reduce anesthetic drug consumption and postoperative analgesia requirements in several types of surgery. Optimal post-operative pain control is necessary for early mobilization, improved respiratory function, and deep venous thrombosis. Administration of multimodal analgesics could limit the excessive use of systemic opioid analgesia especially (morphine), which has a high rate of postoperative side effects as sedation, respiratory depression, ileus, nausea, vomiting, constipation, urine retention, and itching. Therefore, medications and adjuvant drugs reducing the need for opioids have become widely used as parts of multimodal analgesia. Post-operative pain management begins with pre-operative planning and formulating a pain management plan that is tailored to an individual patient's liver function, respiratory and coagulation status, comorbidities and extent of resection.

Anesthetic technique:

Patients will be premedicated with tablet of alprazolam 0.25 mg the night before and 2 hours before surgery. Upon arrival in operating room usual monitoring will be established including heart rate, blood pressure, electrocardiogram (ECG),and temperature. After induction of anesthesia, an arterial line will be inserted for continuous monitoring of blood pressure and frequent blood gas analysis. End-tidal carbon dioxide (capnography) will be attached. General anesthesia will be administered using propofol 2 mg/kg, morphine 0.1 mg/kg and atracurium besylate 0.5 mg/kg followed by oral endotracheal intubation. Maintenance of general anesthesia with a mixture of isoflurane and 50% oxygen in air, morphine 2 mg/ h, mechanical ventilation will be adjusted to keep arterial oxygen saturation < 95 % and end-tidal carbon dioxide between 35 and 40 mmHg. Atracurium (0.15 mg/kg) will be administered every 30 min.

Baseline intravenous infusion rate of lactated ringers solution will be set at (6ml/ kg/h) in both groups, additional solution will be infused if required. Magnesium sulfate infusion and anesthetic agents will be discontinued at the end of operation. The postoperative residual neuromuscular blockade will be reversed by using neostigmine 0.04 mg/kg and atropine 0.02 mg/kg. Then the patient will be extubated and transferred to the post-anesthesia care unit (PACU) for 1-hour observation.

Statistical analysis:

Statistical analysis will be done using Statistical Package for Social Sciences (SPSS) version 19 for Windows software. Data will be collected from all patients during and after anesthesia. Descriptive statistics (mean, standard deviation, or median and ranges) will be calculated. Comparative statistics between the two groups will be applied. Unpaired t-test will be used to compare the mean values between the two groups. The Kolmogorov-Smirnov test will be implemented to check the normality of continuous data distribution (P ≤ 0.05) Mann-Whitney-U test will be used to compare diﬀerence between the two groups for non-parametric variables (e.g.VAS). While the Chi-square test will be used to compare the categorical variables between both groups. The significant result will be considered when P value was less than (0.05).

Sample size calculations of this trial will be done upon the following assumption, α = 0.05 β = 0.2, effect size will be =0.7.The effect size is calculated by using G*Power software version 3.1.9.2 (Institute of Experimental Psychology, Heinrich Heine University, Dusseldorf, German) and the authors found that 25 patients in each group have a power of 80% and plan to recruit 30 patients per group to account for possible dropout.

ELIGIBILITY:
Inclusion Criteria:

* Age (18-50).
* American Society of Anesthesiology (ASA) physical state I or II.
* Normal serum electrolytes.

Exclusion Criteria:

* Impaired hepatic or renal functions.
* Various degree of heart block.
* Hypertension
* Diabetes
* Myopathy or any neurological disorder.
* History of long term opioid use
* Patients treated with calcium channel blockers
* Patients with known allergy to drug used.
* Pregnant woman
* Obesity (Body Mass Index > 30).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-05-08 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Morphine consumption | 24 hours after operation
  in mg

SECONDARY OUTCOMES:
Mean arterial pressure | 1 minute before induction
  in mm mercury by invasive blood pressure
Heart rate | 1 minute before induction
  in beat per minute by electrocardiogram
Mean arterial pressure | 30 seconds before intubation
  in mm mercury by invasive blood pressure
Heart rate | 30 seconds before intubation
  in beat per minute by electrocardiogram
Mean arterial pressure | 5 minutes after beginning of surgery
  in mm mercury by invasive blood pressure
Heart rate | 5 minutes after beginning of surgery
  in beat per minute by electrocardiogram
Mean arterial pressure | 15 minutes after beginning of surgery
  in mm mercury by invasive blood pressure
Heart rate | 15 minutes after beginning of surgery
  in beat per minute by electrocardiogram
Mean arterial pressure | 30 minutes after beginning of surgery
  in mm mercury by invasive blood pressure
Heart rate | 30 minutes after beginning of surgery
  in beat per minute by electrocardiogram
Mean arterial pressure | 60 minutes after beginning of surgery
  in mm mercury by invasive blood pressure
Heart rate | 60 minutes after beginning of surgery
  in beat per minute by electrocardiogram
Mean arterial pressure | 120 minutes after beginning of surgery
  in mm mercury by invasive blood pressure
Heart rate | 120 minutes after beginning of surgery
  in beat per minute by electrocardiogram
Mean arterial pressure | 30 minutes after end of surgery
  in mm mercury by invasive blood pressure
Heart rate | 30 minutes after end of surgery
  in beat per minute by electrocardiogram
Morphine consumption | 30 minutes after end of surgery
  in milligram
Visual Analog Scale | 30 minutes after end of surgery
  Pain score which starting from 0:no pain to 10:Worst pain
Assessment of sedation | 30 minutes after end of surgery
  By 5-point sedation Ramsay score where 5:aroused only by shaking 4:difficult response to verbal 3:mostly sleeping but easily aroused 2:drowsy 1:awake
Mean arterial pressure | 4 hours after end of surgery
  in mm mercury by invasive blood pressure
Heart rate | 4 hours after end of surgery
  in beat per minute by electrocardiogram
Morphine consumption | 4 hours after end of surgery
  in milligram
Visual Analog Scale | 4 hours after end of surgery
  Pain score which starting from 0:no pain to 10:Worst pain
Assessment of sedation | 4 hours after end of surgery
  By 5-point sedation Ramsay score where 5:aroused only by shaking 4:difficult response to verbal 3:mostly sleeping but easily aroused 2:drowsy 1:awake
Mean arterial pressure | 24 hours after end of surgery
  in mm mercury by invasive blood pressure
Heart rate | 24 hours after end of surgery
  in beat per minute by electrocardiogram
Morphine consumption | 24 hours after end of surgery
  in milligram
Visual Analog Scale | 24 hours after end of surgery
  Pain score which starting from 0:no pain to 10:Worst pain
Assessment of sedation | 24 hours after end of surgery
  By 5-point sedation Ramsay score where 5:aroused only by shaking 4:difficult response to verbal 3:mostly sleeping but easily aroused 2:drowsy 1:awake
Mean arterial pressure | 48 hours after end of surgery
  in mm mercury by invasive blood pressure
Heart rate | 48 hours after end of surgery
  in beat per minute by electrocardiogram
Morphine consumption | 48 hours after end of surgery
  in milligram
Visual Analog Scale | 48 hours after end of surgery
  Pain score which starting from 0:no pain to 10:Worst pain
Assessment of sedation | 48 hours after end of surgery
  By 5-point sedation Ramsay score where 5:aroused only by shaking 4:difficult response to verbal 3:mostly sleeping but easily aroused 2:drowsy 1:awake
Patient satisfaction level | 48 hours after end of surgery
  By 5-point scale where 1: very unsatisfactory 2:unsatisfactory 3:neutral 4:satisfactory 5:Excellent
Blood serum magnesium concentration | 12 hours before operation
  from venous blood sample in mg/dl
Blood serum magnesium concentration | 15 minutes after operation
  from venous blood sample in mg/dl
Interleukin 6 level in blood | 24 hours after operation
  inflammatory mediator measured from venous blood sample
Interleukin 8 level in blood | 24 hours after operation
  inflammatory mediator measured from venous blood sample
Tumor necrosis factor alpha level in blood | 24 hours after operation
  inflammatory mediator measured from venous blood sample
Incidence of shivering | 48 hours after operation
  as opioid related side effect
Incidence of nausea | 48 hours after operation
  as opioid related side effect
Incidence of vomiting | 48 hours after operation
  as opioid related side effect
Incidence of respiratory depression | 48 hours after operation
  as opioid related side effect
Incidence of somnolence | 48 hours after operation
  as opioid related side effect
Incidence of oversedation | 48 hours after operation
  as opioid related side effect
Incidence of itching | 48 hours after operation
  as opioid related side effect
Incidence of constipation | 48 hours after operation
  as opioid related side effect
Incidence of paralytic ileus | 48 hours after operation
  as opioid related side effect

OTHER OUTCOMES:
Age | 1 hour before operation once patient is recruited
  in years
Height | 1 hour before operation once patient is recruited
  in meters
Weight | 1 hour before operation once patient is recruited
  in kilogram
body mass index | 1 hour before operation once patient is recruited
  kilogram/meter square
Surgery duration | 1 minute after operation
  in hours
Anesthesia duration | 1 minute after withdrawal of all anesthetics
  in hours from time of induction to withdrawal of all anesthetics

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa S Elhamamsy, MD, Study Chair — Faculty of medicine, Fayoum University; Ahmed M Yassin, MD, Study Director — Faculty of medicine, Beni-suef University; Abeer S Goda, MD, Study Director — Faculty of medicine, Fayoum University; Hany M Yassin, MD, Principal Investigator — Faculty of medicine, Fayoum University
Locations (1):
- Sheikh Zayed hospital, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gucyetmez B, Atalan HK, Aslan S, Yazar S, Polat KY. Effects of Intraoperative Magnesium Sulfate Administration on Postoperative Tramadol Requirement in Liver Transplantation: A Prospective, Double-Blind Study. Transplant Proc. 2016 Oct;48(8):2742-2746. doi: 10.1016/j.transproceed.2016.08.033. PMID 27788811
- [Background] Demiroglu M, Un C, Ornek DH, Kici O, Yildirim AE, Horasanli E, Baskan S, Fikir E, Gamli M, Dikmen B. The Effect of Systemic and Regional Use of Magnesium Sulfate on Postoperative Tramadol Consumption in Lumbar Disc Surgery. Biomed Res Int. 2016;2016:3216246. doi: 10.1155/2016/3216246. Epub 2016 Jan 28. PMID 27022607
- [Background] Sousa AM, Rosado GM, Neto Jde S, Guimaraes GM, Ashmawi HA. Magnesium sulfate improves postoperative analgesia in laparoscopic gynecologic surgeries: a double-blind randomized controlled trial. J Clin Anesth. 2016 Nov;34:379-84. doi: 10.1016/j.jclinane.2016.05.006. Epub 2016 Jun 5. PMID 27687417
- [Background] Yassin HM, Abd Elmoneim AT, El Moutaz H. The Analgesic Efficiency of Ultrasound-Guided Rectus Sheath Analgesia Compared with Low Thoracic Epidural Analgesia After Elective Abdominal Surgery with a Midline Incision: A Prospective Randomized Controlled Trial. Anesth Pain Med. 2017 Jun 10;7(3):e14244. doi: 10.5812/aapm.14244. eCollection 2017 Jun. PMID 28856110
- [Background] Karbasy SH, Derakhshan P. Effects of opium addiction on level of sensory block in spinal anesthesia with bupivacaine for lower abdomen and limb surgery: a case-control study. Anesth Pain Med. 2014 Nov 26;4(5):e21571. doi: 10.5812/aapm.21571. eCollection 2014 Dec. PMID 25798378